CLINICAL TRIAL: NCT05912621
Title: Tirzepatide: Reversal of Lipotoxicity and Adipose Tissue Dysfunction in Humans With Overweight/Obesity
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Tracey McLaughlin, Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 70131
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Obesity; Overweight and Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — Tirzepatide

STUDY DESIGN:
Intervention Model Description: 204 patients with BMI 27-39.9 kg/m2 and fasting plasma glucose < 126 mg/dL will be screened to enroll 68 (to complete 60) who will be randomized 1:1 (computer generated randomization with blocking by sex and BMI category (27-29.9, 30-34.9, 35-39.9 kg/m2) to tirzepatide or dietary weight loss for 22 wks. Individuals with BMI 27-29.9 kg/m2 must have an additional cardiovascular risk factor or weight-related comorbidity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 2.5 mg (up to 15 mg) Tirzepatide (Experimental): Patients assigned to tirzepatide will undergo dose titration starting with 2.5 mg per day with an increase every four weeks if tolerated by nausea. During the first 6 weeks, weight loss must be matched with the dietary weight loss arm at 0.6 kg/week. Participants will be seen every two weeks to review diet and physical activity, evaluate tolerability/side effects, and obtain morning weight. If weight loss is greater than 0.6 kg/week, recommendations to increase caloric intake will be made through the week 6 visits that repeat baseline testings (biopsy, metabolic tests, and regional fat scans). After the 6th week, weight loss can occur naturally without any restrictions (no further matching to the dietary weight loss group is required). Starting at week 8 the visits are decreased to every 4 weeks. Biopsies, metabolic tests, and regional fat scans are completed at baseline, week 6, and end of study (week 22).
  Interventions: Drug: Tirzepatide
- Diet-controlled (No Intervention): The group assigned to dietary weight loss will undergo intensive dietary counseling with initial 3 day food diary evaluation followed by specific dietary recommendations that include macronutrient balanced, healthful and calorie-restricted diet, weekly dietitian visits, alternating between video and in person, use of a mobile app for food logging, weekly weights at home and biweekly weights, and review of these data by the study dietitian who will give individualized feedback at the weekly visits in order to attain targeted weight loss of 0.6 kg per week. The goal is to match weight loss in the tirzepatide and diet groups for the first six weeks. Any residual differences in weight loss at 6 weeks will be adjusted statistically. At six weeks all baseline tests (biopsy, metabolic tests, and regional fat scans) will be repeated, after which no further attempts for matching for weight loss will occur. At the end of the study (week 22), all baseline testing will occur again.

INTERVENTIONS:
Drug: Tirzepatide — Tirzepatide dose is titrated up by 2.5 mg every four weeks as per below, starting with 2.5 mg weekly and maxing out at 15 mg.
  Other Names: Mounjaro
  Arms: 2.5 mg (up to 15 mg) Tirzepatide

SUMMARY:
Obesity, affecting 40% of US adults and costing 173b annually, represents a significant health care burden (1). It is associated with increased risk for multiple chronic diseases including hypertension, type 2 diabetes (T2D), cardiovascular disease, and NAFLD, as well as cancer, osteoarthritis, and obstructive sleep apnea. The investigators plan to test the hypothesis that tirzepatide, a dual GLP/GIP agonist, improves metabolic health (insulin resistance and regional fat distribution and cardiovascular risk profile) not only by inducing weight loss via GLP1-agonism, but also via beneficial cellular and molecular changes in adipose tissue, given that GIP binds receptors in human fat cells. Based on studies in mice showing that GIP alone or tirzepitide treatment decreases inflammation, increases lipid buffering (fat storage in the fat cells instead of releasing it into the bloodstream), and improves glucose homeostasis. The investigators believe that the GIP component of tirzepatide will make fat cells healthier and reverse lipotoxicity, which is one of the mechanisms by which obesity leads to insulin resistance, disordered regional fat distribution, and type 2 diabetes. To date, the effect of dual GLP1 and GIP agonist treatment on adipose tissue has not been evaluated in humans. Given the existing but limited data, dual GIP/GLP-1 agonist treatment in obese humans with metabolic risk factors is an attractive pharmacologic candidate that would lead to both weight loss and healthier fat, potentially offering uniquely powerful synergistic clinical benefits. It is thus of tremendous importance to define the biological effects of dual-agonist treatment on human adipose tissue structure and function, as well as related improvements in regional fat distribution and systemic adipose and muscle insulin sensitivity. In this study, the investigators will randomize overweight (with risk factors) or obese nondiabetic individuals to hypocaloric diet or tirzepatide for 22 weeks with matched weight loss for the first 6 weeks. The investigators will quantify insulin resistance, fat and lean mass, including regional fat distribution, and changes in adipose tissue (needle biopsy from abdominal fat tissue) to see if tirzepatide effects differ from dietary weight loss.

DETAILED DESCRIPTION:
All participants will come to the Stanford University campus for their baseline, week 6, and week 22 (end of study) tests. Prior to starting the assigned intervention, all participants will undergo a supervised (by study dietitian) week of weight maintenance, followed by baseline tests including insulin resistance test (SSPG), Standardized Meal Tolerance Test (for hormone and metabolite profiles), oral glucose tolerance test (OGTT), DXA and MRI scans (to quantify total, regional, and intrahepatic fat), and a subcutaneous periumbilical adipose tissue needle biopsy. Following baseline testing, participants begin tirzepatide vs diet. weight loss will be aggressive for the first six weeks with diet to match the tirzepatide weight loss that is expected. After week 6 weight loss will occur naturally on both without matching. Patients will see the dietitian and coordinator every two weeks to review diet and physical activity, and evaluate tolerability/side effects, and obtain morning weight at Stanford. The metabolic tests, regional fat scans, and biopsy will be repeated at week 6 and week 22.

ELIGIBILITY:
Inclusion Criteria:

* nondiabetic as defined by fasting plasma glucose < 126 mg/dL while off all glucose lowering medications
* BMI 27-39.9 kg/m2. Individuals with obesity (BMI 30-39.9 kg/m2) are not required to have an additional risk factor but those who are overweight (27-29.9 kg/m2) must have at least one weight-related factor as follows: hypertension defined as physician-diagnosed and taking antihypertensive medication or SBP> 130 or DBP > 80 mm Hg; dyslipidemia defined as physician diagnosed and taking medication or LDL > 160 mg/dL, TG > 150 mg/dL, HDL < 50 or < 40 mg/dL for women and men, respectively; prediabetes defined as fasting glucose 100-125 mg/dL off all antidiabetic or diabetogenic medications, physician diagnosed obstructive sleep apnea, non-alcoholic fatty liver disease, history of gallstones, and osteoarthritis.
* Age 18-70
* Pre and postmenopausal women will be eligible and details of last menstrual period and/or hormone replacement collected for statistical adjustment and formal testing for effect modification.

Exclusion Criteria:

* prior bariatric surgery or liposuction
* unstable body weight defined as self-reported weight change >2 kg over the past 6 weeks
* unstable hypertension (defined as BP >160/100 mm Hg)
* major organ disease
* chronic inflammatory conditions
* pregnancy/lactation
* active malignancy undergoing treatment
* use (current or within the past three months) of diabetogenic or weight loss medications, including GLP1 analogs
* active eating or psychiatric disorder
* heavy alcohol use (>2 drinks/day for women and > 3 drinks/day for men) will be excluded

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Change in Adipocyte Size | Baseline and Week 22
  Using a multisizer, we will identify the size and distribution changes of fat cells from baseline to the end of the weight loss period to compare between tirzepatide administration and dietary restriction group
Change in Adipocyte Fat Storage Capacity | Baseline and Week 22
  Using a Oil Red O and rtPCR, we will identify the fat storage capacity of fat cells from baseline to the end of the weight loss period to compare between tirzepatide administration and dietary restriction group
Assess changes in Regional Fat | Baseline, week 6, and week 22
  Using a DXA scan, we will measure the percentages of total, upper, lower, truncal, peripheral, and subcutaneous fat and compare it at baseline, 6 weeks, and 22 weeks for each participant
Change from baseline on the 2-stage Steady State Plasma Glucose test | Baseline, week 6, and week 22
  Compare direct measurement of insulin sensitivity after baseline, week 6, and week 22

CONTACTS AND LOCATIONS:
Overall Officials: Tracey McLaughlin, MD, Principal Investigator — Stanford School of Medicine
Locations (1):
- Clinical and Translational Research Unit, Palo Alto, California, United States